CLINICAL TRIAL: NCT02377141
Title: Early Use of Transjugular Intrahepatic Portosystemic Shunt (TIPSS) in Patients With Cirrhosis and Variceal Bleeding
Brief Title: Early Use of TIPSS in Patients With Cirrhosis and Variceal Bleeding
Acronym: EarlyTIPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 81135
Record Dates: First submitted 2015-02-05; First posted 2015-03-03 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Liver Cirrhosis; Variceal Haemorrhage
Keywords: Oesophageal Variceal Bleed; TIPSS; Endoscopic Variceal Band Ligation; Decompensated Liver Disease
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Variceal Band Ligation (EVBL) (Active Comparator): Participants in this group will receive standard medical care consisting of vasoactive drugs (Terlipressin 2mg QDS (where there are no contraindications e.g. severe ischaemic heart disease), antibiotics, and entry into a variceal banding programme (in-patient or out-patient).
  Interventions: Procedure: Endoscopic Variceal Band Ligation
- Early TIPSS (Active Comparator): For those randomized to early TIPSS the Transjugular Intrahepatic Porto-Systemic Stent Shunt (TIPSS) procedure will be performed within 72 hours (and preferably within the first 24 hours) after initial endoscopy. Vasoactive drugs will be continued until the TIPSS is performed and antibiotics continued for 5-7 days.
  Interventions: Procedure: Endoscopic Variceal Band Ligation; Procedure: Transjugular Intrahepatic Porto-Systemic Stent Shunt

INTERVENTIONS:
Procedure: Endoscopic Variceal Band Ligation — Standard care: Endoscopic application of rubber bands to varices (swollen veins) in the oesophagus this is repeated on 4-5 occasions until the varices are eradicated.
  Other Names: Endosopic banding,; Banding
Procedure: Transjugular Intrahepatic Porto-Systemic Stent Shunt — Within 72 hours of the initial endoscopy to apply bands to the bleeding varices the patient undergoes a Transjugular Intrahepatic Porto-Systemic Stent Shunt (TIPSS) procedure. Under x-ray guidance a shunt is created in the liver between the hepatic vein and portal vein via a catheter introduced via the jugular vein. It may require a check once or twice per year to ensure it remains patent.
  Other Names: TIPSS; TIPS
  Arms: Early TIPSS

SUMMARY:
Gastro-oesophageal varices (swollen veins in the gullet and stomach) are present in 50% of patients with liver cirrhosis and are its most serious complication as their rupture results in potentially life threatening bleeding. Bleeding from these veins occurs in up to one third of patients with varices. This is associated with 20% mortality at 6 weeks.

In the event of bleeding from these veins the current UK guidelines recommend certain drugs followed by early endoscopic treatment with variceal band ligation (rubber bands placed over the veins to stop them bleeding). The use of a shunt inside the liver ("TIPSS" transjugular intrahepatic portosystemic shunt) is largely reserved for cases of uncontrolled bleeding from these swollen veins. A recent randomised multicenter study carried out by Garcia Pagan and colleagues reported improved survival with early TIPSS in patients with bleeding from these swollen veins in advanced liver disease. From these guideline international guidelines now recommend consideration of early TIPSS for all high-risk patients presenting with variceal bleeding. This practice clearly has significant cost implications. To validate the findings a further randomised control trial is needed.

This is a multi-center parallel-group randomized controlled trial. Both hospitals taking part in the trial will have a TIPSS service. Patients who consent to enter the trial will be randomized to either: (1) Endoscopic treatment (standard care) or (2) early TIPSS.

Potential participants will be all patients with a diagnosis of liver cirrhosis presenting with an acute variceal bleed to a participating hospital who do not fulfill an exclusion criteria. All causes of cirrhosis will be included.

Participants will be reviewed during their regular hepatology clinic appointments at their respective hospitals on 3 occasions over a one-year period.

DETAILED DESCRIPTION:
Background and Rationale for the Study

Gastro-oesophageal varices are present in 50% of patients with cirrhosis [2] and are the most serious complication of portal hypertension as their rupture results in potentially life threatening variceal haemorrhage with overall mortality rates historically reported as 30-50% [3]. Although mortality can be up to 40% at 6 weeks, it can be up to 70% at one year [2]. With the generally improved management of critically ill cirrhotic patients, together with vasoactive therapy and new endoscopic techniques for managing variceal haemorrhage, overall mortality has reduced, with one centre in Europe showing a reduction from 42% in 1980 to 14% in 2000 [4]. 60-80% of patients who bleed from varices will re-bleed if not treated [5-8], and the risk of re-bleeding is greatest in the first 10 days [1,9], during which 50% of those who are going to re-bleed, do so. The risk of re-bleeding gradually falls over the first month when an additional 10% re-bleed [7, 8]; the risk after the first six weeks then plateaus out.

Despite the advent of endoscopic therapies and early pharmacological therapies, re-bleeding rates are still higher early on, with factors predictive of early re-bleeding /treatment failure at 5 days including: active bleeding at index endoscopy; severity of liver disease (Child-Pugh class); severity of bleed; and severity of portal hypertension [1, 10]. Hepatic Venous Pressure Gradient (HVPG) is one of the best predictors of identifying those who will re-bleed. After an index variceal bleed, a reduction of HVPG to less than 12mmHg or by at least 20%, reduces the risk of re-bleeding from 46-65% to 0.13% [11]. HVPG measurement is usually limited to specialist centres.

The early use of TIPSS has been explored in two studies [1,12]. The first [12] categorised patients presenting with a variceal bleed to be either high or low risk of re-bleeding determined by their HVPG. Those with an HVPG greater or equal to 20mmHg went on to receive an early TIPSS and had an improved outcome compared with those treated medically. However, the results must be interpreted with caution, as the medical management was not current standard of care.

A further study investigating the use of early TIPSS for variceal haemorrhage was carried out by Garcia-Pagan and colleagues [1]. This landmark study selected patients for early TIPSS (within 3 days) determined by Child-Pugh score. Participants, who had Child's B or C cirrhosis and on-going bleeding, progressed to early use of TIPSS (with an e-PFTE-covered stent). The results of this trial demonstrated a significant reduction in the failure to control bleeding and re-bleeding with no increase in the risk of hepatic encephalopathy. The study also demonstrated a significant survival benefit with early TIPSS at all time points. There were, however, several features of this study that raised concern.

Firstly recruitment was prolonged (3 years) to recruit 63 patients via 9 centres, with a high exclusion rate (296 patients excluded). The second concern featured the inclusion of patients with ongoing bleeding following index endoscopy. This might arguably be termed a rescue TIPSS and although no studies have been done in this area it is intuitive to suggest that survival would be improved if haemostasis has not been achieved. Thirdly, survival at 1 year with early TIPSS was extremely high (86% vs. 61% in the medical management group). For patients with Child's C cirrhosis presenting with variceal bleeding this survival rate is remarkable.

These two studies [1, 12] of the early use of TIPSS for variceal haemorrhage are the first in portal hypertension to show a mortality benefit. As such these demand action. Either the management of variceal bleeding in patients with advanced cirrhosis must change or, given the concerns regarding the study design and the significant cost implications, these results need to be further validated.

STUDY DESIGN This is a multi-centre, open-label, parallel-group, randomised control trial. Both hospitals taking part in the trial will have a 24-hour TIPSS service. Potential participants will be all patients with a diagnosis of liver cirrhosis presenting with variceal haemorrhage to a participating hospital who do not fulfil an exclusion criteria. Potential participants will be identified by the gastroenterology team responsible for the patient care. Patients and their relatives will be approached by a nominated registrar, or consultant, identified in the ethics application or delegation log. Patients will be followed up for one year and will be reviewed on three occasions. Patients who consent to enter the trial will be randomized to either: (1) EVBL ("standard care") arm or (2) early TIPSS arm.

FOLLOW UP During their regular Hepatology follow-ups, patients will be reviewed at 6 weeks, 6 months, and 12 months, which is the end of the study. TIPSS patency will be checked at 6 months and 1 year as per current standard protocol. All patients will be followed up until death or the end of the study, whichever is first.

IDENTIFYING PARTICIPANTS Potential participants will be all patients with a diagnosis of liver cirrhosis presenting with an acute variceal haemorrhage to a participating hospital who do not fulfil an exclusion criteria. All aetiologies of cirrhosis (including cryptogenic and where the aetiology is yet to be established) will be included. Potential participants will be identified by the gastroenterology team responsible for the patient. The consultant responsible for the care of each patient will determine whether the identified patients are suitable and may be approached.

OBTAINING CONSENT If patients are alert and able to give informed consent then they will be issued with a patient information sheet and consent sought from the patient. Patients and their next of kin will have sufficient time usually 3 hours or more, from the index endoscopy to consent to inclusion in the study.

Patients with liver disease may have fluctuating conscious level and may lack capacity due to hepatic encephalopathy. Potential participants who lack capacity will be included in the study. Here capacity will be assessed by the consenting clinician at the time of taking consent. A further consent will be sought from those patients who regain capacity.

RANDOMISATION This study will involve simple 1:1 randomisation. Randomisation will be done using a web-based randomisation programme that will be available 24 hours a day to both study centres.

STUDY ASSESSMENT Participants will attend the gastroenterology/hepatology clinics at their respective hospital on three occasions over a one-year period. If participants are in hospital at the time of a scheduled visit then they will either be assessed whilst inpatient or at the programmed visit as an outpatient. The programme visits are: 6 Weeks, 6 Months and 1 year.

SAMPLE SIZE CALCULATION Given that we are validating results of the Garcia Pagan study, we have powered the study using the results that they observed. We wish to find a difference in survival between the two trial arms. Garcia Pagan observed 14% and 39% deaths in the two trial arms. We calculate that we would need 48 patients per group. This is from a 2-sided log-rank test, with alpha=0.05, and a power of 80%, allowing 4 extra patients per group to allow for drop out and non-compliance.

ELIGIBILITY:
Inclusion Criteria:

* An acute oesophageal variceal bleed with haemostasis following initial endoscopy.
* A diagnosis of liver cirrhosis
* Childs-Pugh score ≥8

Exclusion Criteria:

* Inability to control bleeding at index endoscopy (this is a "rescue TIPSS")
* Previous portosystemic shunt or TIPSS
* Bleeding from isolated gastric or ectopic varices
* Known portal vein thrombosis precluding TIPSS
* Active cancer including hepatocellular carcinoma
* Age less than 18 or more than 75
* Clinically significant encephalopathy causing recurrent hospital admissions
* Pregnant at time of index endoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Survival | One Year
  Patient survival at 1 year

SECONDARY OUTCOMES:
Survival | 6 weeks
  Patient survival at 6 weeks
Liver Transplant-free survival | To liver transplant (time not defined)
  For patients eligible for a liver transplant the time from study entry to transplantation will be noted.
Rate of early re-bleeding | Within 6 weeks
  Recurrent bleeding from oesophageal varices
Rate of late re-bleeding | 6 weeks to 1 year
  Recurrent bleeding from oesophageal varices
The development of hepatic encephalopathy | Anytime within the year
  Time to development of hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Hayes, MD PhD, Study Chair — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow

REFERENCES:
- [Background] Garcia-Pagan JC, Caca K, Bureau C, Laleman W, Appenrodt B, Luca A, Abraldes JG, Nevens F, Vinel JP, Mossner J, Bosch J; Early TIPS (Transjugular Intrahepatic Portosystemic Shunt) Cooperative Study Group. Early use of TIPS in patients with cirrhosis and variceal bleeding. N Engl J Med. 2010 Jun 24;362(25):2370-9. doi: 10.1056/NEJMoa0910102. PMID 20573925
- [Background] de Franchis R; Baveno V Faculty. Revising consensus in portal hypertension: report of the Baveno V consensus workshop on methodology of diagnosis and therapy in portal hypertension. J Hepatol. 2010 Oct;53(4):762-8. doi: 10.1016/j.jhep.2010.06.004. Epub 2010 Jun 27. No abstract available. PMID 20638742
- [Background] D'Amico G, Pagliaro L, Bosch J. The treatment of portal hypertension: a meta-analytic review. Hepatology. 1995 Jul;22(1):332-54. doi: 10.1002/hep.1840220145. No abstract available. PMID 7601427
- [Background] Carbonell N, Pauwels A, Serfaty L, Fourdan O, Levy VG, Poupon R. Improved survival after variceal bleeding in patients with cirrhosis over the past two decades. Hepatology. 2004 Sep;40(3):652-9. doi: 10.1002/hep.20339. PMID 15349904
- [Background] D'Amico G. The role of vasoactive drugs in the treatment of oesophageal varices. Expert Opin Pharmacother. 2004 Feb;5(2):349-60. doi: 10.1517/eoph.5.2.349.26486. PMID 14996631
- [Background] de Franchis R. Evolving consensus in portal hypertension. Report of the Baveno IV consensus workshop on methodology of diagnosis and therapy in portal hypertension. J Hepatol. 2005 Jul;43(1):167-76. doi: 10.1016/j.jhep.2005.05.009. No abstract available. PMID 15925423
- [Background] Graham DY, Smith JL. The course of patients after variceal hemorrhage. Gastroenterology. 1981 Apr;80(4):800-9. PMID 6970703
- [Background] D'Amico G, De Franchis R; Cooperative Study Group. Upper digestive bleeding in cirrhosis. Post-therapeutic outcome and prognostic indicators. Hepatology. 2003 Sep;38(3):599-612. doi: 10.1053/jhep.2003.50385. PMID 12939586
- [Background] Matsumoto A, Hamamoto N, Nomura T, Hongou Y, Arisaka Y, Morikawa H, Hirata I, Katsu K. Balloon-occluded retrograde transvenous obliteration of high risk gastric fundal varices. Am J Gastroenterol. 1999 Mar;94(3):643-9. doi: 10.1111/j.1572-0241.1999.00928.x. PMID 10086645
- [Background] Bambha K, Kim WR, Pedersen R, Bida JP, Kremers WK, Kamath PS. Predictors of early re-bleeding and mortality after acute variceal haemorrhage in patients with cirrhosis. Gut. 2008 Jun;57(6):814-20. doi: 10.1136/gut.2007.137489. Epub 2008 Feb 4. PMID 18250126
- [Background] Bosch J, Garcia-Pagan JC. Prevention of variceal rebleeding. Lancet. 2003 Mar 15;361(9361):952-4. doi: 10.1016/S0140-6736(03)12778-X. PMID 12648985
- [Background] Monescillo A, Martinez-Lagares F, Ruiz-del-Arbol L, Sierra A, Guevara C, Jimenez E, Marrero JM, Buceta E, Sanchez J, Castellot A, Penate M, Cruz A, Pena E. Influence of portal hypertension and its early decompression by TIPS placement on the outcome of variceal bleeding. Hepatology. 2004 Oct;40(4):793-801. doi: 10.1002/hep.20386. PMID 15382120
- [Derived] Dunne PDJ, Sinha R, Stanley AJ, Lachlan N, Ireland H, Shams A, Kasthuri R, Forrest EH, Hayes PC. Randomised clinical trial: standard of care versus early-transjugular intrahepatic porto-systemic shunt (TIPSS) in patients with cirrhosis and oesophageal variceal bleeding. Aliment Pharmacol Ther. 2020 Jul;52(1):98-106. doi: 10.1111/apt.15797. Epub 2020 May 26. PMID 32452561